CLINICAL TRIAL: NCT00591201
Title: Efficacy, Safety, and Tolerability of Infliximab (Remicade; Schering-Plough) in Juvenile Spondyloarthropathies: a Three-Month, Randomized, Double-Blind, Placebo-Controlled Trial and 52-Week Open Extension.
Brief Title: Efficacy, Safety, and Tolerability Study of Infliximab in Juvenile Spondyloarthropathies
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hospital General de Mexico (Other Government)
Collaborators: Schering-Plough (Industry)
Responsible Party: Rubén Burgos-Vargas/Professor of Medicine, Medical Doctor., Hospital General de México and Universidad Nacional Autónoma de México
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HGMREUMA.001.2007; DIC/02/404-B/02/036
Record Dates: First submitted 2007-12-31; First posted 2008-01-11 (Estimated); Last update posted 2008-01-17 (Estimated); Status verified 2007-12

CONDITIONS: Spondylarthropathies
Keywords: Spondylarthritis; TNF; Infliximab; Ankylosing spondylitis; Juvenile SpA; Juvenile arthritis
MeSH Terms: conditions — Spondylarthropathies; Spondylarthritis; Spondylitis, Ankylosing; Arthritis, Juvenile | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Infliximab
  Interventions: Drug: infliximab
- B (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: infliximab — Infliximab 5mg/kg diluted in 250 ml of isotonic solution of sodium chloride will be administered by the intravenous route on weeks 0, 2, 6, 12, 18, 24, 30, 36, 42, and 48.
  Other Names: remicade
  Arms: A
Drug: Placebo — Placebo -powder diluted in 250 ml of isotonic solution of sodium chloride- will be administered on weeks 0, 2 and 6.
  Arms: B

SUMMARY:
Tumor necrosis factor (TNF) alpha is a pro-inflammatory cytokine playing a significant role in the pathogenesis of the spondyloarthropathies (SpA). Infliximab is a TNF alpha blocking monoclonal antibody efficacious and safe as treatment of adult-onset SpA.

In this study we will try to demonstrate that infliximab administered at 5mg/kg to patients with juvenile onset SpA over a period of 12 weeks will have more efficacy than placebo and that it will be well tolerated. At the end of this phase, patients will go into a 52-week open extension to demonstrate sustained efficacy, safety, and tolerability of infliximab We will include 34 patients with juvenile onset SpA unresponsive to standard treatment. Efficacy will be assessed by counting the number of actively inflamed joints and a number of other parameters.

DETAILED DESCRIPTION:
Background Tumor necrosis factor (TNF) alpha is a pro-inflammatory cytokine playing a significant role in the pathogenesis of the spondyloarthropathies (SpA). Infliximab is a TNF alpha blocking monoclonal antibody efficacious and safe as treatment of adult-onset SpA.

Hypothesis Infliximab will reduce the number of joints with active arthritis and improve additional parameters of disease activity and functioning more significantly than placebo over 12 weeks. Infliximab will demonstrate sustained efficacy and its administration will be safe and well tolerated over 52 weeks.

Objectives To demonstrate superior clinical efficacy with infliximab administered at 5mg/kg compared with placebo, in juvenile onset SpA over a period of 12 weeks. To demonstrate sustained efficacy, safety, and tolerability of infliximab at 5 mg/kg over 52 weeks.

Study Design This is a two-phase study. First phase: 12-week, randomized, double-blind, placebo-controlled period to evaluate efficacy, safety, and tolerability of infliximab 5 mg/kg.

Thirty-four patients allocated and randomized to infliximab 5 mg/kg or placebo. Randomization: restricted by blocks of four and by stratification in two diagnostic categories (undifferentiated SpA and ankylosing spondylitis). Efficacy analysis: change of the primary efficacy measure and secondary measures on weeks 2, 6, and 12, and any visit of discontinuation compared to week 0 and compared to changes in the placebo group.

Patients completing the 1st phase and those discontinued due to lack of efficacy after week 6 will continue into the 2nd phase to complete a total of 52 weeks. The 2nd open-phase will demonstrate the sustained efficacy, safety, and tolerability of infliximab along 52 weeks (weeks 12, 18, 24, 30, 36, 42 and 48). Efficacy analysis will focus on the change of the primary efficacy measurement and secondary measures on each scheduled visits- and any discontinuation visit compared to week 0.

Safety Evaluation Safety evaluations will included a search for clinical serious and non-serious adverse events; blood cytology, hepatic function tests, blood chemistry, urinanalysis, antinuclear antibodies by immunofluorescence, anti-DNA antibodies, rheumatoid factor, and chest X-rays.

Statistical Analysis The primary analysis will follow the "intention to treat" model. The data of patients who have been prematurely discontinued from the study- since V2.0- will be included in the primary analysis. The comparison between infliximab and placebo will be sequential.

Double-blind phase: step-down analysis; changes from baseline will be computed from a time-weighted average of the responses across weeks 2, 4, and 6 -and any discontinuation visit. 95% confidence intervals to evaluate the magnitude of the difference between infliximab and placebo will be used.

Open phase: mean changes from baseline on the time weighted average of responses over the whole length of the study.

Statistical tests: parametric and non parametric to evaluate the inter and intragroupal differences; ANCOVA, Mann Whitney, Wilcoxon, t of student and x2.

Sample size: 17 patients per group, plus 2 patients per group because of loss, supposes an improvement in the study group of 60% to 90%, with a confidence level of 95% to 99% (two tails test) and a power of 80% to 90%, with improvement in the control group of only 10%. The basis of such calculations is indirect because there are no data about juvenile SpA; yet, data on adults treated with infliximab and children and teenagers treated with sulfasalazine compared to placebo exist.

Budget The project and protocol are the result of the initiative of the investigators who are the intellectual proprietaries of it. Schering Plough, owner of the patent of Infliximab (Remicade; Schering Plough), has accepted to finance the project.

ELIGIBILITY:
Inclusion Criteria:

* Ages less tha 16 years at symptoms onset and less than 18 years at entry
* SpA diagnoses (ESSG criteria)
* Active arthritis at least 2 peripheral joints
* Pressure tenderness at least 3 peripheral entheses
* Pain intensity of 40 mm in an analogue visual scale (VAS)
* Lack of response to NSAID, sulfasalazine or methotrexate
* Serum HCG-beta levels congruent with no pregnancy
* Use of double-barrier contraceptive methods
* History of BCG vaccination
* Capacity to understand the study and follow protocol instructions
* Written and signed consent letter.

Exclusion criteria:

* Pregnancy and lactation
* Mental disability
* Functional class IV
* Psoriasis, reactive arthritis or inflammatory bowel disease
* Infectious, neoplastic, metabolic, hepatic, hematological, vascular, cardiopulmonary or renal active diseases
* Opportunistic infectious
* Active tuberculosis
* Significant laboratory tests abnormalities
* Current prednisone dose of more than 10 mg/day;
* Intraarticular/muscular/venous glucocorticoids
* Previous use of Infliximab or etanercept, pentoxyphylline, thalidomide, or anti-CD4 antibodies
* Allergy or hypersensitivity to infliximab
* Significant drug changes within one month before screening
* Use of recreational drugs/illicit substances.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2002-06; Primary Completion 2007-06 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Number of joints with active arthritis. | 12 weeks

SECONDARY OUTCOMES:
Number of tender entheses; patient assessment of pain; patient/parent assessment of well being; investigator assessments of disease activity and health status; childhood health assessment questionnaire; and C reactive protein. Safety issues | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Burgos-Vargas, MD, Principal Investigator — Rheumatologist, Hospital General de México/Professor of Medicine, Universidad Nacional Autónoma de México
Locations (1):
- Servicio de Reumatología, Hospital General de México, Mexico City, Mexico City, Mexico